CLINICAL TRIAL: NCT06530797
Title: A Multicenter Real-World Cohort Study of Adebrelimab Injection in the Treatment of Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Ren Shengxiang, Prof., Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: OBU-SH-SCLC-RWS-001
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Keywords: Extensive-stage small cell lung cancer (ES-SCLC); Adebrelimab
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-line treatment for advanced stage: Any first-line regiment including Adebrelimab for advanced stage ES-SCLC
  Interventions: Drug: First-line Adebrelimab regiment for advanced stage ES-SCLC
- Second-line and beyond for advanced stage: Any Second- or later-line and regiment including Adebrelimab for advanced stage ES-SCLC
  Interventions: Drug: Second-line and beyond Adebrelimab regiment for advanced stage ES-SCLC

INTERVENTIONS:
Drug: First-line Adebrelimab regiment for advanced stage ES-SCLC — First-line Adebrelimab in any regiment for advanced stage ES-SCLC
  Groups: First-line treatment for advanced stage
Drug: Second-line and beyond Adebrelimab regiment for advanced stage ES-SCLC — Second-line and beyond Adebrelimab in any regiment for advanced stage ES-SCLC
  Groups: Second-line and beyond for advanced stage

SUMMARY:
The purpose of this observational study is to evaluate the safety and efficacy of Adebrelimab Injection in extensive-stage small cell lung cancer (ES-SCLC) under real-world conditions. Specifically, the study aims to assess the treatment of Adebrelimab Injection across various subgroups of ES-SCLC patients. The goal is to provide information on treatment patterns and effectiveness in real-life settings, explore potential predictive or prognostic biomarkers, and preliminarily evaluate the pharmacoeconomic indicators of Adebrelimab Injection treatment for extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
This trial is a multicenter, non-interventional real-world study aimed at evaluating the safety and efficacy of Adebrelimab in the treatment of extensive-stage small cell lung cancer (ES-SCLC). The study plans to enroll 2000 patients with extensive-stage small cell lung cancer, collecting relevant information such as demographics, medical history, treatment regimens including Adebrelimab, clinical outcomes, and adverse events.

Patients who have already decided to receive Adebrelimab treatment before enrollment will be categorized into one of the following two cohorts based on their disease stage and prior treatments:

Cohort 1: First-line treatment for advanced stage Cohort 2: Second-line and beyond for advanced stage

The Adebrelimab-containing treatment regimen for each patient will be assessed and selected by the investigator, and some treatment regimens are provided in this protocol for reference. After patients discontinue Adebrelimab treatment, they will be followed up until death, loss to follow-up, withdrawal of informed consent/voluntary withdrawal, or study termination/closure, whichever occurs first.

As this is an observational study, treatments, procedures, visits, and examinations are based on the routine clinical experience of the attending physicians. The examinations listed in the protocol are recommended or for reference, with no mandatory requirements. The primary source of data for this study will be patients' routine medical records. During the period of Adebrelimab treatment, data on the administration regimen, routine examinations, adverse events, concomitant medications, and efficacy evaluations will be collected.

When patients permanently discontinue Adebrelimab treatment for any reason (including but not limited to disease progression, intolerable toxicity, patient request, etc.), the reasons for discontinuation, adverse events/serious adverse events (up to 90 days after the last dose of Adebrelimab), the time of radiographic disease progression (if not the reason for discontinuation), subsequent anti-tumor treatments, and survival follow-up data will be collected.

This study will explore potential predictive or prognostic biomarkers for ES-SCLC, so patients are requested to provide 10 tumor tissue slides whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for inclusion in this study:

  1. Voluntarily sign the informed consent form and agree to participate in the study.
  2. Histopathologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC).
  3. Age ≥ 18 years.
  4. Determined by the investigator to be eligible for Adebrelimab treatment.

Exclusion Criteria:

* Patients with any of the following conditions are not eligible for inclusion in this study:

  1. Evidence of being a pregnant or lactating female.
  2. Currently receiving treatment as part of a blinded study protocol.
  3. Any other condition that the investigator deems unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For some adverse reactions with an incidence as low as 0.25%, further observation in a larger population in the real world is needed. Using NCSS PASS 21 software (LLC. Kaysville, Utah, USA, ncss.com/software/pass), it was calculated that approximately 2000 patients need to be observed in this study to ensure a confidence of no less than 99% in successfully observing at least one case of an adverse reaction with an incidence as low as 0.25%.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety (The occurrence of ≥3 grade AEs) | From August 2024, patients will be followed up for 90 days after the last use of Adebrelimab
  The occurrence of ≥3 grade AEs

SECONDARY OUTCOMES:
PFS | Up to 2 years. From date of enrollment until the date of first documented progression, assessed up to 2 years.
  Progression free survival from Adebrelimab treatment
OS | Up to 2 years. From date of enrollment until the date of death from any cause, assessed up to 2 years.
  Overall survival from Adebrelimab treatment
DoR | Up to 2 years. From date of enrollment until the date of first documented progression, assessed up to 2 years.
  Duration of response of Adebrelimab treatment
ORR | Up to 2 years. From date of enrollment until the date of first documented progression, assessed up to 2 years.
  Objective response rate of Adebrelimab treatment
DCR | Up to 2 years. From date of enrollment until the date of first documented progression, assessed up to 2 years.
  Disease control rate of Adebrelimab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shengxiang Ren, MD., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956
- [Result] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287